CLINICAL TRIAL: NCT00960752
Title: Activation of pDCs at the Tumor and Vaccine Site With a Toll Like Receptor (TLR) Agonist
Brief Title: Tumor and Vaccine Site With a Toll Like Receptor (TLR) Agonist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0416; NCI-2011-02363 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Melanoma
Keywords: gp100 peptide; MAGE-3 peptide; R848; Resiquimod; Toll Like Receptor; TLR; T-cells; Tumor; Metastatic; Lesions; Injection Site
MeSH Terms: conditions — Melanoma; Neoplasms; Neoplasm Metastasis | interventions — gp100 Melanoma Antigen; g209-2M melanoma peptide; resiquimod; MAGEA3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: gp100 and MAGE-3 + R848 (Active Comparator): 1 ml of gp100 peptide vaccine and 1 ml of MAGE-3 peptide vaccine daily for 8 weeks with R848 Gel applied to gp100 injection site immediately. Injections given intradermally and subcutaneously at 2 separate sites in separate extremities. Half of each dose given one way, and half given the other way. Vaccines given on the same day. Participant receives a total of 4 injections each week.
  After 8 weeks, if participant has melanoma lesions, R848 applied to half of the lesions on body for 16 weeks.
  Interventions: Drug: gp100; Drug: R848 gel; Drug: MAGE-3
- Group 2: gp100 and MAGE-3 (Active Comparator): 1 ml of gp100 peptide vaccine and 1 ml of MAGE-3 peptide vaccine daily for 8 weeks. Injections given intradermally and subcutaneously at 2 separate sites in separate extremities. Half of each dose given one way, and half given the other way. Vaccines given on the same day. Participant receives a total of 4 injections each week.
  After 8 weeks, if participant has melanoma lesions, R848 applied to half of the lesions on body for 16 weeks.
  Interventions: Drug: gp100; Drug: MAGE-3
- Group 3-Metastatic Melanoma: gp100 + MAGE-3 + R848 (Active Comparator): 1 ml of gp100 peptide vaccine and 1 ml of MAGE-3 peptide vaccine daily for 8 weeks with R848 Gel applied to gp100 injection site immediately. Injections given intradermally and subcutaneously at 2 separate sites in separate extremities. Half of each dose given one way, and half given the other way. Vaccines given on the same day. Participant receives a total of 4 injections each week.
  After 8 weeks, if participant has melanoma lesions, R848 applied to half of the lesions on body for 16 weeks.
  Interventions: Drug: gp100; Drug: R848 gel; Drug: MAGE-3

INTERVENTIONS:
Drug: gp100 — 1 ml of gp100 peptide vaccine: 0.5 ml administered intradermally and the other 0.5 ml subcutaneously in the same extremity weekly (every 7 days +/- 2 days) for 8 weeks.
  Other Names: gp100 peptide; g209-2M
Drug: R848 gel — Applied to the gp100 vaccine injection site immediately following the injection, allowed to air dry for 30 minutes then covered with gauze dressing.
  Other Names: Resiquimod
  Arms: Group 1: gp100 and MAGE-3 + R848; Group 3-Metastatic Melanoma: gp100 + MAGE-3 + R848
Drug: MAGE-3 — 1 ml of MAGE-3 peptide vaccine: 0.5 ml administered intradermally and the other 0.5 ml subcutaneously in the same extremity weekly (every 7 days +/- 2 days) for 8 weeks.
  Other Names: MAGE-3 peptide

SUMMARY:
The goal of this clinical research study is to learn if the vaccines, gp100(g209-2M), and MAGE-3, when given in combination with resiquimod (R848), can help to stimulate the immune system against melanoma.

DETAILED DESCRIPTION:
The Study Drug/Vaccines:

Resiquimod (R848) is designed to increase the production of antigen-specific T-cells, to activate immune cells, and to increase T-cells going into the tumor, which may cause the tumor cells to die.

gp100(g209-2M) and MAGE-3 are vaccines designed to stimulate immune cells, also called T-cells, which may help the immune system to recognize and kill melanoma cells.

Study Groups:

If you are found to be eligible to take part in this study, and you have metastatic melanoma, you will be assigned to Group 3. If you have had the melanoma removed and want to be treated to try to keep it from coming back, you will be randomly assigned (as in the flip of a coin) to Group 1 or 2.

* If you are in Group 1, you will receive the vaccines gp100(g209-2M) and MAGE-3 and R848 for 8 weeks. After 8 weeks, if you have melanoma lesions, you will apply R848 to half of the lesions on your body for 16 weeks.
* If you are in Group 2, you will receive only the vaccines (gp100(g209-2M) and MAGE-3) only for 8 weeks. After 8 weeks, if you have melanoma lesions, you will apply R848 to half of the lesions on your body for 16 weeks.
* If you are in Group 3, you will receive the vaccines gp100(g209-2M) and MAGE-3 and R848 for 8 weeks. After 8 weeks, if you have melanoma lesions, you will apply R848 to half of the lesions on your body for 16 weeks.

After 8 weeks, if you no longer have melanoma lesions, you will have completed the study treatment.

Study Drug/Vaccine Administration:

Once a week for 8 weeks, you will receive the vaccines, gp100(g209-2M) and MAGE-3, intradermally (through a needle into your skin) and subcutaneously (through a needle under your skin) at 2 separate sites in separate extremities. Half of each dose will be given one way, and half given the other way. These vaccines will also be given on the same day. You will receive a total of 4 injections each week.

If you are in Group 1, every time you have the vaccine injection, R848 will be applied as a gel over the gp100(g209-2M) injection site. The R848 gel will be allowed to air dry for 30 minutes and then covered with a gauze dressing which remain on overnight.

After 8 weeks, for participants with melanoma lesions, 2 times a week for 16 weeks, you will apply the R848 gel to half of the lesions on your body. You will be given written instructions and a "hands-on" demonstration on how to apply the gel. You will also be given a worksheet to help you with applying the gel.

Study Visits:

One day after your first dose of vaccine (Day 2), you will have a punch biopsy of the vaccine injection site to check your immune system. A punch biopsy is when a hollow instrument that is used to remove a small coin-shaped sample of tissue.

At Week 2, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be recorded.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Blood (about 4 tablespoons) will be drawn to study your immune response to the vaccine combinations.
* You will have a punch biopsy of the injection site to check your immune system the day after the vaccine is given.

Every 4 weeks, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be recorded.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Blood (about 4 tablespoons) will be drawn to study your immune response to the vaccine combinations.

Every 8 weeks, for participants with metastatic disease, the following tests and procedures will be performed:

* You will have CT or PET/CT scans of the chest, abdomen, and pelvis to check the status of the disease.
* The tumors will be measured and photographed. Your private areas will be covered (as much as possible), and a picture of your face will not be taken unless there are tumors on your face.
* If the doctor thinks it is necessary, the tumors will be measured by CT scan.
* If the doctor thinks it is needed, you will have an MRI/CT of the brain to check the status of the disease.

The day after you first start the gel (Week 8), you will have 2 punch tumor biopsies to check your immune system. One biopsy will be of a lesion with the R848 and one without, if it is available. For participants without disease, the study will be completed and your follow-up will be decided by your doctor.

At Week 0 (before vaccine is started), after treatment at Week 8 (+/- 1 week)., and Week 16 (+/- 1 week), white blood cells will be collected by leukapheresis to test for antibodies. If you have the leukapheresis, blood (about 2 teaspoons) will be drawn as well. If you do not have leukapheresis, blood (about 4 tablespoons) will be drawn instead.

The leukapheresis procedure is research-related and would not be performed as standard of care if you were not on study. Blood for the leukapheresis will be taken through a needle in a vein in one of your arms. A solution will be added to keep your blood from clotting while it goes through the machine that collects and removes white blood cells from your blood. The remaining blood is returned to you through a needle in a vein of your other arm. This is may take up to 3-4 hours. Although several pints of blood will go through the machine, only about 1/2 a pint (1 cup) will be in the machine at any time. If you cannot have a needle in your vein, this blood will be removed thorough a central venous catheter (CVC). A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. You will be given another informed consent document to sign, which describes the risks of the CVC and the care involved.

Length of Study:

You will continue to receive treatment for up to 4 6 months, as long as you may benefit from the study and are responding to the gel. You will be taken off study if the disease gets worse or you experience any intolerable side effects. If you are in the group without disease, you will not receive the study treatment.

Follow-Up:

All three groups will be called 1 time a month for 12 months after coming off the study drugs to check on the status of the disease.

This is an investigational study. The study drugs/vaccines gp100(g209-2M), MAGE-3, and R848 are not FDA approved or commercially available. At this time, they are only being used in research.

Up to 71 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. HLA-A*0201 positive (to enable immunization with the HLA class I restricted gp100(g209-2M) peptide). Stage IIB or IIC patients will be enrolled after review and approval by the PI. (a tool to determine the projected survival at 5 years, like, but not limited to, the nomogram at www.melanomaprognosis.org. If the projected survival is less than 50% at 5 years, then the patient is considered for enrollment. This is with the recognition that the adjuvant, if effective offers a significant impact in that group of stage II patients.)
2. Patients >/= 18 years old with histologically documented metastatic melanoma with a. (Metastatic disease cohort) Measurable disease, stage IIIB, IIIC (in transit lesions with or without nodal metastases) that includes lesions accessible for biopsies or IV M1B b. (Adjuvant cohort) subjects who are NED and stage III or IV. This includes patients with stage IV disease resected to NED. Stage IIB or IIC patients will be enrolled after review and approval by the PI.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
4. At least 2 biopsiable easily accessible cutaneous and subcutaneous lesions in patients in the metastatic disease cohort
5. White Blood Count (WBC) >/= 3000/mm^3 (part 1 & 2)
6. Platelet count >/= 90,000/mm^3 (part 1 & 2)
7. Serum alanine aminotransferase (ALT) and Aspartate Aminotransferase (AST) </= 3 X upper limit of normal (ULN) (part 1 & 2)
8. Total bilirubin </= 2 X ULN, except for patients with Gilbert's syndrome who must have a total bilirubin less than 3.0 mg/dl Total bilirubin </= 2 X ULN, except for patients with Gilbert's syndrome who must have a total bilirubin less than 3.0 mg/dl (part 1 & 2)
9. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities.)
10. Negative pregnancy test for women of childbearing potential (WOCBP) A WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses at any time in the preceding 12 consecutive months)
11. Patients of both gender must practice a barrier method of birth control while participating in this trial.

Exclusion Criteria:

1. Active autoimmune disease requiring active therapy with any form of steroid or immunosuppressive therapy or a documented history of any of the following: inflammatory bowel disease; regional enteritis; systemic lupus erythematosis; Sjogren's syndrome; inflammatory neurologic disorder such as multiple sclerosis; or any immune mediated disease that can cause life-threatening symptoms or severe organ/tissue damage in the opinion of the principle investigator.
2. Concurrent systemic or inhaled steroid therapy
3. Any form of active primary or secondary immunodeficiency
4. Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, thyroid cancer (except anaplastic) or any cancer from which the patient has been disease-free for 2 years
5. History of immunization with gp100(g209-2M)
6. Active systemic infections requiring intravenous antibiotics
7. Women who are breastfeeding
8. Prior systemic therapy, radiation therapy or intracavitary surgery (intra-thoracic, intra-abdominal or intracranial) within 28 days of starting study treatment.
9. Patients on chronic anticoagulation such as Aspirin, Plavix, or Coumadin who cannot have anticoagulation held for procedures are not eligible due to the need for leukapheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-05-20 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Davies, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 participants enrolled on study, 1 participant screen failure, 1 participant stopped prematurely due to toxicity.
Groups:
- Group 1: GP100 and MAGE-3 + R848; Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848: 1 ml of gp100 peptide vaccine and 1 ml of MAGE-3 peptide vaccine daily for 8 weeks with R848 Gel applied to gp100 injection site immediately.
- Group 2: GP100 and MAGE-3: 1 ml of gp100 peptide vaccine and 1 ml of MAGE-3 peptide vaccine daily for 8 weeks.
Period: Overall Study
Arm/Group | Group 1: GP100 and MAGE-3 + R848 | Group 2: GP100 and MAGE-3 | Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848
Started | 13 | 13 | 19
Completed | 13 | 13 | 17
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Progression | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: GP100 and MAGE-3 + R848 | Group 2: GP100 and MAGE-3 | Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848 | Total
Number analyzed (Participants) | 13 | 13 | 19 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 4 | 24
  >=65 years | 2 | 4 | 15 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 13
  Male | 8 | 9 | 15 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 12 | 13 | 18 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 13 | 19 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 19 | 45

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Immune Responses of Vaccine+R848 to Vaccine Alone
Description: T-cell response to gp100(g209-2M) +/- MAGE3 measured at 8 weeks using a tetramer/multimer assay measured by flow cytometry. Based on the number of gp100(g209-2M) +/- MAGE3 T-cells measured, categorized as either immune responders or immune non-responders. T-cell response to the gp100(g209-2M) + /- MAGE3 peptide in each participant defined as ≥0.1% gp100(g209-2M) tetramer+ cells in the CD8+ T-cell population or ≥0.1% MAGE3 multimer cells in the CD4+ T-cell population.
Time Frame: 8 weeks
Population: The original PI is no longer in the institution. Due to the absence of the original PI is no longer in the institution and the data is unavailable. The analysis for the primary outcome measure the comparison of immune responses of vaccine+R848 to vaccine alone is not available. All efforts were made to retrieve data.
Arm/Group | Group 1: GP100 and MAGE-3 + R848 | Group 2: GP100 and MAGE-3 | Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Composite of Immune Cell Infiltration for pDCs, mDCs, and NK Cells in Tumor Biopsy Samples
Description: Differences determined in each of these parameters between the pretreatment and post-treatment samples for each of the biopsied lesions for each participant.
Time Frame: 8 weeks
Population: The original PI is no longer in the institution. Due to the absence of the original PI is no longer in the institution and the data is not available. The analysis for the secondary outcome measure the composite of Immune Cell Infiltration for pDCs, mDCs, and NK cells in Tumor Biopsy Samples data is unavailable .All efforts were made to retrieve data.
Arm/Group | Group 1: GP100 and MAGE-3 + R848 | Group 2: GP100 and MAGE-3 | Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: every 2 weeks through Week 4, then every 4 weeks during the vaccination treatment, up to 8 weeks
Arm/Group | Group 1: GP100 and MAGE-3 + R848 | Group 2: GP100 and MAGE-3 | Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 2/19
Other Adverse Events (participants affected / at risk) | 13/13 | 9/13 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: GP100 and MAGE-3 + R848 (N=13) | Group 2: GP100 and MAGE-3 (N=13) | Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848 (N=19)
Platelet Count Decreased (Blood and lymphatic system disorders) | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: GP100 and MAGE-3 + R848 (N=13) | Group 2: GP100 and MAGE-3 (N=13) | Group 3-Metastatic Melanoma: GP100 + MAGE-3 + R848 (N=19)
Injection Site Reaction (General disorders) | 13 | 8 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 9 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 5 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Rhinitis infective (Infections and infestations) | 3 | 2 | 2
Chills (General disorders) | 0 | 0 | 6
Dizziness (Nervous system disorders) | 4 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT00960752/Prot_SAP_000.pdf